CLINICAL TRIAL: NCT00918255
Title: A Phase 2 Multicenter Study of the Safety and Efficacy of Adalimumab in Subjects With Moderate to Severe Chronic Hidradenitis Suppurativa
Brief Title: Study of Adalimumab in Subjects With Moderate to Severe Chronic Hidradenitis Suppurativa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Martin Okun, Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-467; 2008-004587-38 (EudraCT Number)
Record Dates: First submitted 2009-04-30; First posted 2009-06-11 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis Suppurativa; Adalimumab; Nodule; Abscess; Fistula; Physicians Global Assessment; Hurley Stage; Sartorius Scale
MeSH Terms: conditions — Hidradenitis Suppurativa; Abscess; Fistula | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Adalimumab 40 mg qwk (Experimental): Initial dose of adalimumab 160 mg at Week 0, adalimumab 80 mg at Week 2, followed by 40 mg weekly (qwk) starting at Week 4 through Week 15.
  Interventions: Biological: adalimumab
- Adalimumab 40 mg eow (Experimental): Initial dose of adalimumab 80 mg at Week 0, followed by adalimumab 40 mg eow (every other week) starting at Week 1 through Week 15.
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator): Matching placebo for adalimumab, administered weekly starting at Week 0 through Week 15.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: adalimumab — Subcutaneous injection using prefilled syringe containing adalimumab 40 mg in 0.8 milliliters
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 40 mg eow; Adalimumab 40 mg qwk
Drug: Placebo — Subcutaneous injection using prefilled syringe containing 0.8 milliliters
  Arms: Placebo

SUMMARY:
This study will investigate how well adalimumab works in people with hidradenitis suppurativa (HS) in the short and long term.

DETAILED DESCRIPTION:
This Phase 2 randomized, double-blind, placebo-controlled multicenter study consists of 2 treatment periods: a 16-week double-blind, placebo-controlled period (Period 1: Weeks 0 through the end of Week 15) followed by a 36-week open-label period (Period 2: Weeks 16 through 52). Participants are randomized in a 1:1:1 ratio based on Hurley Stage as stratification factor to receive adalimumab 40 mg every week (qwk), adalimumab 40 mg every other week (eow), or matching placebo during Period 1. During Period 2, participants receive open-label adalimumab 40 mg eow with the option to escalate to 40 mg weekly dosing at Week 28 or Week 31 if the participant has a Physician's Global Assessment of moderate disease or worse (score of greater than or equal to 3). The primary objective of the study is to determine the clinical efficacy and safety of participants with moderate to severe chronic hidradenitis suppurativa (HS) after 16 weeks of treatment. The secondary objective is to evaluate the maintenance of efficacy and continued safety of adalimumab for an additional 36 weeks of treatment. (Note: Hurley Stage is a classification system for skin involvement that is largely based on the presence and extent of abscess formation accompanied by scarring and sinus tracts. Hurley Stages are I [abscess formation without scarring and sinus tracts], II [widely separated recurrent abscesses with scarring and sinus tracts], and III [multiple interconnected abscesses and sinus tracts across entire area]. Randomization in this study was performed using stratification by Hurley Stage [III versus (I or II).) At the present time, Period 1 double-blind data only is provided; additional information will be provided when analysis of open-label Period 2 is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stable, moderate to severe hidradenitis suppurativa
* Negative Chest X-ray and PPD test at Screening. If participant has had a past ulcerative reaction to PPD placement and/or chest X-ray consistent with prior tuberculosis exposure, the participant must initiate, or have documented completion of, a course of anti-tuberculosis therapy.
* Ability to administer subcutaneous injections
* General good health otherwise

Exclusion Criteria:

* Prior anti-TNF therapy
* Unstable antibiotic therapy for HS
* Required medication washouts for other HS treatments
* Prior exposure to Tysabri® (natalizumab);
* Recent infection requiring treatment
* Significant medical events or conditions that may put patients at risk for participation
* Female subjects who are pregnant or breast-feeding or considering becoming pregnant during the study;
* History of cancer, except successfully treated skin cancer
* Recent history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Okun, MD, PhD, Study Director — Abbott
Locations (26):
- United States (20):
  - Site Ref # / Investigator 19062, Birmingham, Alabama
  - Site Ref # / Investigator 18201, Bakerfield, California
  - Site Ref # / Investigator 18467, Los Angeles, California
  - Site Ref # / Investigator 18207, San Diego, California
  - Site Ref # / Investigator 18204, Miami, Florida
  - Site Ref # / Investigator 18209, Atlanta, Georgia
  - Site Ref # / Investigator 18202, Skokie, Illinois
  - Site Ref # / Investigator 18211, Evansville, Indiana
  - Site Ref # / Investigator 18203, Boston, Massachusetts
  - Site Ref # / Investigator 18210, Boston, Massachusetts
  - Site Ref # / Investigator 18461, St Louis, Missouri
  - Site Ref # / Investigator 18466, Omaha, Nebraska
  - Site Ref # / Investigator 19141, New York, New York
  - Site Ref # / Investigator 18208, New York, New York
  - Site Ref # / Investigator 19001, Winston-Salem, North Carolina
  - Site Ref # / Investigator 18981, Hershey, Pennsylvania
  - Site Ref # / Investigator 18464, Philadelphia, Pennsylvania
  - Site Ref # / Investigator 19061, Dallas, Texas
  - Site Ref # / Investigator 18463, San Antonio, Texas
  - Site Ref # / Investigator 18206, Norfolk, Virginia
- Denmark (2):
  - Site Ref # / Investigator 18683, Copenhagen NV
  - Site Ref # / Investigator 18684, Roskilde
- Germany (2):
  - Site Ref # / Investigator 18471, Dessau
  - Site Ref # / Investigator 18469, Kiel
- Netherlands (2):
  - Site Ref # / Investigator 18470, Amsterdam
  - Site Ref # / Investigator 18468, Rotterdam

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Scheinfeld N, Sundaram M, Teixeira H, Gu Y, Okun M. Reduction in pain scores and improvement in depressive symptoms in patients with hidradenitis suppurativa treated with adalimumab in a phase 2, randomized, placebo-controlled trial. Dermatol Online J. 2016 Mar 16;22(3):13030/qt38x5922j. PMID 27136622
- [Derived] Kimball AB, Kerdel F, Adams D, Mrowietz U, Gelfand JM, Gniadecki R, Prens EP, Schlessinger J, Zouboulis CC, van der Zee HH, Rosenfeld M, Mulani P, Gu Y, Paulson S, Okun M, Jemec GB. Adalimumab for the treatment of moderate to severe Hidradenitis suppurativa: a parallel randomized trial. Ann Intern Med. 2012 Dec 18;157(12):846-55. doi: 10.7326/0003-4819-157-12-201212180-00004. PMID 23247938

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab 40 mg Qwk DB: Initial dose of adalimumab 160 mg at Week 0, adalimumab 80 mg at Week 2, followed by 40 mg weekly (qwk) starting at Week 4 through Week 15.
- Adalimumab 40 mg Eow DB: Initial dose of adalimumab 80 mg at Week 0, followed by adalimumab 40 mg eow (every other week) starting at Week 1 through Week 15.
- Placebo DB: Matching placebo for adalimumab, administered weekly starting at Week 0 through Week 15.
Period: Overall Study
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Started | 51 | 52 | 51
Completed | 45 | 52 | 46
Not Completed | 6 | 0 | 5
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Exceeded allowed number of interventions | 0 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Investigator discretion | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adalimumab 40 mg Qwk DB: Loading dose of adalimumab 160 mg at Week 0, adalimumab 80 mg at Week 2, followed by 40 mg weekly (qwk) starting at Week 4 through Week 15.
- Adalimumab 40 mg Eow DB: Loading dose of adalimumab 80 mg at Week 0, followed by adalimumab 40 mg eow (every other week) starting at Week 1 through Week 15.
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB | Total
Number analyzed (Participants) | 51 | 52 | 51 | 154
Age Continuous [Mean (Standard Deviation); unit: years] | 35.1 (10.69) | 36.1 (12.50) | 37.8 (12.10) | 36.3 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 36 | 110
  Male | 15 | 14 | 15 | 44
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 36 | 116
  Europe | 10 | 13 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response at Week 16
Description: Clinical response is defined as a Physician's Global Assessment (PGA) of clear, minimal, or mild (scores of 0, 1, or 2) with a minimum of 2 grades improvement (reduction) from baseline. PGA is a physician's assessment of the severity of disease based on a 6-point scale (score of 0 = clear and 5 = very severe).
Time Frame: Baseline, Week 16
Population: Intent-to-treat analysis with non-responder imputation (participants with missing PGA scores counted as non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
percentage of participants | 17.6 | 9.6 | 3.9
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel — When this initial overall comparison of the 3 treatment groups was significant, pairwise comparisons of each adalimumab dose group versus placebo were performed
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.252, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage

2. Secondary Outcome: Percent Change From Baseline in Number of All Inflammatory Nodules and Plaques at Week 16
Description: Includes inflammatory nodules that are tender, erythematous, and have diameters less than 5 cm and includes plaques that have diameters greater than or equal to 5 cm. Range for percent change is negative infinity to infinity. Negative percent changes from Baseline indicate improvement.
Time Frame: Baseline, Week 16
Population: Population was Intent-to-treat (ITT) and included participants with any inflammatory nodules (defined as tender, erythematous) or plaques at Baseline. Imputation method was Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 49 | 48 | 48
percent change | -50.66 (11.364) | -30.43 (11.452) | -13.66 (11.452)
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.062, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 0.019, ANCOVA; Analyzed using ANCOVA adjusting for Baseline Hurley Stage (I/II vs III)
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.286, ANCOVA; Analyzed using ANCOVA adjusting for Baseline Hurley Stage (I/II vs III)

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 2
Description: as for outcome 1
Time Frame: Baseline, Week 2
Population: Intent-to-treat analysis with non-responder imputation (participants with missing PGA scores counted as non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
percentage of participants | 2.0 | 9.6 | 2.0
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.097, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage

4. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Population: Intent-to-treat analysis with non-responder imputation (participants with missing PGA scores counted as non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
percentage of participants | 11.8 | 5.8 | 2.0
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.044, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 0.051, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.320, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage

5. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Intent-to-treat analysis with non-responder imputation (participants with missing PGA scores counted as non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
percentage of participants | 7.8 | 5.8 | 7.8
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 1.000, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.673, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage

6. Secondary Outcome: Percentage of Participants Achieving Clinical Response at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: Intent-to-treat analysis with non-responder imputation (participants with missing PGA scores counted as non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
percentage of participants | 21.6 | 7.7 | 5.9
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.721, Cochran-Mantel-Haenszel; Analyzed using CMH test stratified by Hurley Stage

7. Secondary Outcome: Change From Baseline in Modified Sartorius Scale at Week 16
Description: The Modified Sartorius Scale reflects changes in hidradenitis suppurative symptoms, namely the number of lesions (abscesses, nodules, and fistulas) and the longest distance between lesions. A total score is derived based on assessments at up to 8 distinct anatomical regions and ranges from 5 to indefinite. Smaller numbers are better scores and indicate less lesion involvement, thus decreases (negative changes) from baseline indicate improvement in severity of disease.
Time Frame: Baseline, Week 16
Population: Population was Intent-to-treat (ITT). Imputation method was Last Observation Carried Forward (LOCF).
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Number analyzed (Participants) | 51 | 52 | 51
scores on a scale | -30.0 (53.82) [-50.0 to -7.0] | -16.0 (82.54) [-47.0 to 0.0] | -7.5 (47.78) [-30.0 to 10.0]
Statistical Analysis 1: Comparison: Adalimumab 40 mg Qwk DB vs Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.045, Van Elteren test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Adalimumab 40 mg Qwk DB vs Placebo DB; Test type: Superiority or Other; p = 0.014, Van Elteren test; Analyzed using Van Elteren test stratified by Hurley Stage
Statistical Analysis 3: Comparison: Adalimumab 40 mg Eow DB vs Placebo DB; Test type: Superiority or Other; p = 0.169, Van Elteren test; Analyzed using Van Elteren test stratified by Hurley Stage

8. Secondary Outcome: Change From Baseline in Modified Sartorius Scale at Week 52
Description: as for outcome 7
Time Frame: Baseline, Week 52
Reporting Status: Not Posted
Measure: unit: scores on a scale

9. Secondary Outcome: Percent Change From Baseline in Number of All Inflammatory Nodules and Plaques at Week 52
Description: as for outcome 2
Time Frame: Baseline, Week 52
Reporting Status: Not Posted
Measure: unit: percent change

ADVERSE EVENTS:
Time Frame: For the 3 treatment groups in Period 1 (Adalimumab 40 mg Qwk, Adalimumab 40 mg Eow, and Placebo): Week 0 up to Week 16. For Open-label adalimumab (Period 2): Week 16 through Week 52 plus 70 days after the last dose.
Description: Assessment and recording of adverse events and serious adverse events was performed by the investigator at each study visit. Information on events that occurred 70-days after the last dose of study drug (Week 52 or early termination) was collected during a follow-up phone call.
Arm/Group | Adalimumab 40 mg Qwk DB | Adalimumab 40 mg Eow DB | Placebo DB
Serious Adverse Events (participants affected / at risk) | 4/51 | 3/52 | 2/51
Other Adverse Events (participants affected / at risk) | 36/51 | 33/52 | 30/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Qwk DB (N=51) | Adalimumab 40 mg Eow DB (N=52) | Placebo DB (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 1 | 0 | 0
Genital infection bacterial (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1 | 0
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg Qwk DB (N=51) | Adalimumab 40 mg Eow DB (N=52) | Placebo DB (N=51)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3
Fatigue (General disorders) | 3 | 2 | 2
Folliculitis (Infections and infestations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 6 | 7 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Headache (Nervous system disorders) | 8 | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 4 | 6 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Injection site pruritus (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2
Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 2
Herpes simplex (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 2
Blood cholesterol increased (Investigations) | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.